CLINICAL TRIAL: NCT04734392
Title: Reducing Pacemaker Implantation After TAVR With Modified Implantation Technique
Acronym: MIDAS - ULM
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Dr. Dominik Buckert, PD Dr. Dominik Buckert, MD, University of Ulm
Other Study IDs: 01/2021
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: PM Implantation After TAVR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Historical cohort 2019 + 2020
- Cohort B: Prospective study cohort 2020 + 2021 (TAVR implantation according new IFU)
  Interventions: Procedure: TAVR

INTERVENTIONS:
Procedure: TAVR — TAVR implantation in cusp overlay technique
  Groups: Cohort B

SUMMARY:
Hypothesis of the study is that a modified and improved implantation protocol (regarding membranous septum length and implantation depth) will decrease the need for permanent pacemaker stimulation follow TAVR-procedures.

DETAILED DESCRIPTION:
Project objectives or hypothesis Hypothesis of the study is that a modified and improved implantation protocol (regarding membranous septum length and implantation depth) will decrease the need for permanent pacemaker stimulation following TAVR-procedures.

Patient profile and sample size The study cohort will comprise of patients referred to transcatheter aortic valve replacement. Patients will be prospectively and consecutively screened and enrolled at a tertiary high-volume center in Germany. TAVR will be performed according to a modified implantation technique regarding membranous septum length. Pacemaker rates will be analyzed and compared to a historical control. Taking into account a contemporary pacemaker rate of 15%, a reduction to 7% will require a sample size of 239 patients per group to achieve statistically significance (Chi-squared test, alpha 0.05, beta 0.80).

Regarding the prospective cohort, interims analysis will be performed after each 10 TAVR procedures. In case a signal towards worse outcomes with the modified implantation technique will be observed, the institutional safety and endpoint adjudication committee will stop further execution of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to TAVR procedure due to severe aortic stenosis

Exclusion Criteria:

* PM-implantation before TAVR
* Valve-in-valve procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study cohort will comprise of patients referred to transcatheter aortic valve replacement. Patients will be prospectively and consecutively screened and enrolled at a tertiary high-volume center in Germany.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Pacemaker implantation rate | Day 5 after TAVR
  Primary endpoint

SECONDARY OUTCOMES:
Extent of paravalvular leak | Day 5 after TAVR
  Secondary endpoint
Number of patients alive | 30 days
  Secondary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Ulm University, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided